CLINICAL TRIAL: NCT06181435
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallelgroup, 3-arm, Multinational, Multicenter Study to Evaluate the Efficacy and Safety of Amlitelimab Monotherapy by Subcutaneous Injection in Participants Aged 12 Years and Older With Moderate-to-severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Efficacy and Safety of Subcutaneous Amlitelimab Monotherapy Compared With Placebo in Participants Aged 12 Years and Older With Moderate-to-severe Atopic Dermatitis (COAST 2)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17560; 2023-506557-38 (Registry Identifier: CTIS); U1111-1275-9665 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Amlitelimab dose 1 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab
- Amlitelimab dose 2 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab
- Placebo (Placebo Comparator): Subcutaneous injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlitelimab — Pharmaceutical form: Injection solution Route of administration: SC injection
  Other Names: SAR445229
  Arms: Amlitelimab dose 1; Amlitelimab dose 2
Drug: Placebo — Pharmaceutical form:
  Injection solution Route of administration: SC injection
  Arms: Placebo

SUMMARY:
This is a parallel group, Phase 3, multinational, multicenter, randomized, double-blind, placebo-controlled, 3-arm monotherapy study for treatment of participants diagnosed with moderate to severe atopic dermatitis (AD), whose disease is not adequately controlled with topical prescription therapies or when those therapies are not advisable.

The purpose of this study is to measure the efficacy and safety of treatment with amlitelimab solution for SC injection compared with placebo in participants with moderate to severe AD aged 12 years and older.

Study details include:

At the end of the treatment period, participants will have an option to enter a separate study: the blinded extension study EFC17600 (ESTUARY).

For participants not entering the blinded extension Study EFC17600 (ESTUARY), the study duration will be up to 44 weeks including a 2 to 4-week screening, a 24-week randomized double-blind period, and a 16-week safety follow-up.

For participants entering the blinded extension Study EFC17600 (ESTUARY), the study duration will be up to 28 weeks including a 2 to 4-week screening and a 24-week randomized double-blind period.

The total treatment duration will be up to 24 weeks. The total number of visits will be up to 10 visits (or 9 visits for those entering the blinded extension study EFC17600 (ESTUARY).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 12 years of age (when signing informed consent form)
* Diagnosis of AD for at least 1 year (defined by the American Academy of Dermatology Consensus Criteria)
* Documented history (within 6 months before screening) of either inadequate response or inadvisability to topical treatments, and/or inadequate response to systemic therapies (within 12 months before screening)
* v-IGA-AD of 3 or 4 at baseline visit
* EASI score of 16 or higher at baseline
* AD involvement of 10% or more of BSA at baseline
* Weekly average of daily PP-NRS of ≥ 4 at baseline visit.
* Able and willing to comply with requested study visits and procedures
* Body weight ≥ 25 kg

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Skin co-morbidity that would adversely affect the ability to undertake AD assessments
* Known history of or suspected significant current immunosuppression
* Any malignancies or history of malignancies prior to baseline (with the exception of non-melanoma skin cancer excised and cured >5 years prior to baseline)
* History of solid organ or stem cell transplant
* Any active or chronic infection including helminthic infection requiring systemic treatment within 4 weeks prior to baseline
* Positive for human immunodeficiency virus (HIV), Hepatitis B or hepatitis C at screening visit
* Having active tuberculosis (TB), latent TB, a history of incompletely treated TB, suspected extrapulmonary TB infection, or who are at high risk of contracting TB
* Having received any of the specified therapy within the specified timeframe(s) prior to the baseline visit
* In the Investigator's opinion, any clinically significant laboratory results or protocol specified laboratory abnormalities at screening
* History of hypersensitivity or allergy to any of the excipients or investigational medicinal product (IMP)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
EU, EU reference countries, and Japan: Proportion of participants with Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points at Week 24 | Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
EU, EU reference countries, and Japan: Proportion of participants reaching 75% reduction from baseline in Eczema Area and Severity Index (EASI) score (EASI-75) at Week 24 | Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
US and US reference countries: Proportion of participants with vIGA-AD of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points at Week 24 | Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).

SECONDARY OUTCOMES:
Proportion of participants reaching EASI-75 at Week 24 (for US and US reference countries only) | Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score.
Proportion of participants with vIGA-AD 0 (clear) or 1 (almost clear) with presence of only barely perceptible erythema (no induration/papulation, no lichenification, no oozing or crusting) and a reduction from baseline of ≥2 points | Baseline to Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants with ≥4-point reduction in weekly average of daily Peak Pruritus-Numerical Rating Scale (PP-NRS) from baseline in participants with baseline weekly average of daily PP-NRS ≥4 | Baseline to Week 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Proportion of participants reaching EASI-75 | Baseline to Week 20
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score.
Proportion of participants with vIGA-AD of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points | Baseline to Week 20
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants with vIGA-AD 0 (clear) | Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants reaching EASI-90 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-90 is 90% reduction from baseline in EASI score.
Proportion of participants reaching EASI-100 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-100 is 100% reduction from baseline in EASI score.
Proportion of participants with PP-NRS 0 or 1 | Baseline to Week 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Change in Dermatology Life Quality Index (DLQI) from baseline in participants with age ≥16 years old | Baseline to Week 24
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Proportion of participants with a reduction in DLQI ≥4 from baseline in participants with age ≥16 years old and with DLQI baseline ≥4 | Baseline to Week 24
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Change in Children Dermatology Life Quality Index (CDLQI) from baseline in participants with age ≥12 to <16 years old | Baseline to Week 24
  The CDLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in children aged 4-<16 years. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Proportion of participants with a reduction in CDLQI ≥6 from baseline in participants with age ≥12 to <16 years old and with CDLQI baseline ≥6 | Baseline to Week 24
  The CDLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in children aged 4-<16 years. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL
Change in Hospital Anxiety Depression Scale (HADS) from baseline | Baseline to Week 24
  The HADS is 14-item questionnaire with two subscales: anxiety & depression. Each subscale (anxiety & depression) ranges 0-21. The total HADS score ranges 0-42 with higher score indicating a poorer state.
Proportion of participants with HADS subscale Anxiety (HADS-A) <8 in participants with baseline HADS-A ≥8 | Baseline to Week 24
  HADS-A score ranges 0-21 with higher score indicating a poorer state.
Proportion of participants with HADS subscale Depression (HADS-D) <8 in participants with HADS-D baseline ≥8 | Baseline to Week 24
  HADS-D score ranges 0-21 with higher score indicating a poorer state.
Absolute change in weekly average of daily Skin Pain-Numerical Rating Scale (SP-NRS) from baseline | Baseline to Week 24
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Proportion of participants with a reduction in weekly average of daily SP-NRS ≥4 from baseline in participants with baseline weekly average of daily SP-NRS ≥4 | Baseline to Week 24
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Absolute change in weekly average of daily Sleep Disturbance-Numerical Rating Scale (SD-NRS) from baseline | Baseline to Week 24
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Proportion of participants with a reduction in weekly average of daily SD-NRS ≥3 from baseline in participants with Baseline weekly average of daily SD-NRS ≥3 | Baseline to Week 24
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Percent change in weekly average of daily SP-NRS from baseline | Baseline to Week 24
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Percent change in weekly average of daily SD-NRS from baseline | Baseline to Week 24
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Percent change in EASI score from baseline | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Percent change in weekly average of daily PP-NRS from baseline | Baseline to Week 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Absolute change in weekly average of daily PP-NRS from baseline | Baseline to Week 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Proportion of participants reaching EASI-50 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-50 is 50% reduction from baseline in EASI score.
Proportion of participants with EASI ≤7 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Change in percent Body Surface Area (BSA) affected by AD from baseline | Baseline to Week 24
Percent change in Scoring Atopic Dermatitis (SCORAD) index from baseline | Baseline to Week 24
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Absolute change in SCORAD index from baseline | Baseline to Week 24
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Proportion of participants with a reduction in SCORAD ≥ 8.7 points from baseline in participants with baseline SCORAD score ≥ 8.7 | Baseline to Week 24
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Change in Patient Oriented Eczema Measure (POEM) from baseline | Baseline to Week 24
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a 5-point scale; 0 (no days) to 4 (every day in the last week). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (very severe). Higher scores indicated more severe disease and poor quality of life.
Proportion of participants with a reduction in POEM ≥4 from baseline in participants with POEM Baseline ≥4 | Baseline to Week 24
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a 5-point scale; 0 (no days) to 4 (every day in the last week). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (very severe). Higher scores indicated more severe disease and poor quality of life.
Proportion of participants with rescue medication use | Baseline to Week 24
Percentage of participants who experience Treatment-Emergent Adverse Events (TEAEs), experience Treatment-Emergent Serious Adverse Events (TESAEs) and/or Treatment- Emergent Adverse Events of Special Interest (AESI) | Baseline to Week 40
Serum amlitelimab concentrations | Baseline to Week 40
Incidence of antidrug antibodies (ADAs) of amlitelimab | Baseline to Week 40

CONTACTS AND LOCATIONS:
Locations (142):
- United States (43):
  - Center for Dermatology and Plastic Surgery- Site Number : 8401119, Scottsdale, Arizona
  - Eclipse Clinical Research- Site Number : 8401158, Tucson, Arizona
  - Torrance Clinical Research- Site Number : 8401027, Lomita, California
  - Dermatology Research Associates - Los Angeles- Site Number : 8401092, Los Angeles, California
  - Allergy & Asthma Associates of Southern California - Mission Viejo- Site Number : 8401079, Mission Viejo, California
  - Cura Clinical Research - Oxnard- Site Number : 8401142, Oxnard, California
  - Clinical Science Institute- Site Number : 8401028, Santa Monica, California
  - University of Connecticut Health Center- Site Number : 8401115, Farmington, Connecticut
  - Pediatric Skin Research- Site Number : 8401198, Coral Gables, Florida
  - Skin Care Research - Hollywood- Site Number : 8401071, Hollywood, Florida
  - Savin Medical Group - Miami- Site Number : 8401085, Miami, Florida
  - Anchor Medical Research- Site Number : 8401300, Miami, Florida
  - Accel Research - Nona Pediatric Center- Site Number : 8401081, Orlando, Florida
  - Nuline Clinical Trial Center- Site Number : 8401161, Pompano Beach, Florida
  - Clinical Research Trials of Florida- Site Number : 8401023, Tampa, Florida
  - AllerVie Clinical Research - Columbus- Site Number : 8401104, Columbus, Georgia
  - First Georgia Physician Group- Site Number : 8401190, Fayetteville, Georgia
  - Access Dermatology- Site Number : 8401296, Bowling Green, Kentucky
  - MedPharmics - Covington- Site Number : 8401137, Covington, Louisiana
  - Care Access Research - Marriottsville- Site Number : 8401126, Marriottsville, Maryland
  - Tufts Medical Center Site Number : 8401201, Boston, Massachusetts
  - University Of Mississippi Medical Center- Site Number : 8401184, Jackson, Mississippi
  - Care Access - Hoboken- Site Number : 8401132, Hoboken, New Jersey
  - University of New Mexico Comprehensive Cancer Center- Site Number : 8401263, Albuquerque, New Mexico
  - OmeraNY- Site Number : 8401156, Brooklyn, New York
  - Equity Medical- Site Number : 8401239, New York, New York
  - Montefiore Medical Center - Moses Campus- Site Number : 8401150, The Bronx, New York
  - Red River Research Partners- Site Number : 8401196, Fargo, North Dakota
  - Bexley Dermatology Research- Site Number : 8401051, Bexley, Ohio
  - Velocity Clinical Research - Springdale- Site Number : 8401153, Cincinnati, Ohio
  - Dermatology Associates of Plymouth Meeting- Site Number : 8401147, Plymouth Meeting, Pennsylvania
  - PEAK Research- Site Number : 8401083, Upper Saint Clair, Pennsylvania
  - Columbia Dermatology & Aesthetics- Site Number : 8401166, Columbia, South Carolina
  - Health Concepts- Site Number : 8401059, Rapid City, South Dakota
  - Arlington Research Center- Site Number : 8401248, Arlington, Texas
  - Derm Texas- Site Number : 8401217, Dallas, Texas
  - Center for Clinical Studies - Houston - Binz Street- Site Number : 8401063, Houston, Texas
  - Prolato Clinical Research Center- Site Number : 8401209, Houston, Texas
  - Sienna Dermatology- Site Number : 8401148, Missouri City, Texas
  - Progressive Clinical Research - San Antonio- Site Number : 8401016, San Antonio, Texas
  - Advanced Research Institute - Odgen- Site Number : 8401057, Ogden, Utah
  - Care Access - Arlington- Site Number : 8401134, Arlington, Virginia
  - Velocity Clinical Research - Hampton- Site Number : 8401154, Hampton, Virginia
- Argentina (9):
  - Investigational Site Number : 0320021, Berazategui, Buenos Aires
  - Investigational Site Number : 0320017, Pilar, Buenos Aires
  - Investigational Site Number : 0320006, Rosario, Santa Fe Province
  - Investigational Site Number : 0320007, Rosario, Santa Fe Province
  - Investigational Site Number : 0320015, Rosario, Santa Fe Province
  - Investigational Site Number : 0320016, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320009, Buenos Aires
- Bulgaria (3):
  - Investigational Site Number : 1002008, Gabrovo
  - Investigational Site Number : 1002004, Pleven
  - Investigational Site Number : 1002005, Sofia
- Chile (5):
  - Investigational Site Number : 1520004, Valdivia, Los Ríos Region
  - Investigational Site Number : 1520013, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520014, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520015, Quillota, Región de Valparaíso
- China (16):
  - Investigational Site Number : 1560004, Beijing
  - Investigational Site Number : 1560030, Beijing
  - Investigational Site Number : 1560022, Chengdu
  - Investigational Site Number : 1560021, Guangzhou
  - Investigational Site Number : 1560025, Guangzhou
  - Investigational Site Number : 1560002, Hangzhou
  - Investigational Site Number : 1560006, Hangzhou
  - Investigational Site Number : 1560029, Hangzhou
  - Investigational Site Number : 1560007, Jinan
  - Investigational Site Number : 1560024, Ningbo
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560005, Shanghai
  - Investigational Site Number : 1560026, Shenyang
  - Investigational Site Number : 1560023, Wenzhou
  - Investigational Site Number : 1560003, Wuxi
  - Investigational Site Number : 1560028, Zhenjiang
- Czechia (5):
  - Investigational Site Number : 2032106, Kutná Hora
  - Investigational Site Number : 2030010, Olomouc
  - Investigational Site Number : 2032104, Ostrava
  - Investigational Site Number : 2030011, Prague
  - Investigational Site Number : 2030006, Prague
- Denmark (3):
  - Investigational Site Number : 2080002, Aalborg
  - Investigational Site Number : 2080001, Aarhus
  - Investigational Site Number : 2080003, Herlev
- Italy (5):
  - Investigational Site Number : 3800018, Rozzano, Milano
  - Investigational Site Number : 3800013, Rome, Roma
  - Investigational Site Number : 3800009, Catania
  - Investigational Site Number : 3800008, Pisa
  - Investigational Site Number : 3800022, Vicenza
- Japan (18):
  - Investigational Site Number : 3920009, Chitose, Hokkaido
  - Investigational Site Number : 3923114, Obihiro, Hokkaido
  - Investigational Site Number : 3920008, Sapporo, Hokkaido
  - Investigational Site Number : 3920006, Kobe, Hyōgo
  - Investigational Site Number : 3920005, Sagamihara, Kanagawa
  - Investigational Site Number : 3923113, Yokohama, Kanagawa
  - Investigational Site Number : 3920010, Miyagi-gun, Miyagi
  - Investigational Site Number : 3920011, Sendai, Miyagi
  - Investigational Site Number : 3923109, Habikino, Osaka
  - Investigational Site Number : 3923110, Sakai, Osaka
  - Investigational Site Number : 3920002, Iruma, Saitama
  - Investigational Site Number : 3923106, Mibu, Tochigi
  - Investigational Site Number : 3920004, Chūō, Tokyo
  - Investigational Site Number : 3923107, Minato, Tokyo
  - Investigational Site Number : 3920001, Tachikawa, Tokyo
  - Investigational Site Number : 3923108, Kagoshima
  - Investigational Site Number : 3923102, Kyoto
  - Investigational Site Number : 3920003, Kyoto
- Mexico (5):
  - Investigational Site Number : 4840011, Monterrey, Nuevo León
  - Investigational Site Number : 4840005, Monterrey, Nuevo León
  - Investigational Site Number : 4840012, Aguascalientes
  - Investigational Site Number : 4840009, Durango
  - Investigational Site Number : 4840003, Veracruz
- Portugal (4):
  - Investigational Site Number : 6200005, Lisbon
  - Investigational Site Number : 6200004, Lisbon
  - Investigational Site Number : 6200001, Lisbon
  - Investigational Site Number : 6200003, Porto
- South Africa (8):
  - Investigational Site Number : 7100004, Boksburg
  - Investigational Site Number : 7100010, Cape Town
  - Investigational Site Number : 7100009, Cape Town
  - Investigational Site Number : 7100012, Durban
  - Investigational Site Number : 7100001, Durban
  - Investigational Site Number : 7100015, Johannesburg
  - Investigational Site Number : 7100007, Johannesburg
  - Investigational Site Number : 7100003, Pretoria
- Spain (4):
  - Investigational Site Number : 7240012, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number : 7240018, Granada
  - Investigational Site Number : 7240029, Madrid
  - Investigational Site Number : 7242503, Madrid
- Sweden (2):
  - Investigational Site Number : 7520006, Älvsjö
  - Investigational Site Number : 7520001, Örebro
- Turkey (Türkiye) (7):
  - Investigational Site Number : 7920001, Antalya
  - Investigational Site Number : 7920005, Istanbul
  - Investigational Site Number : 7920006, Istanbul
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920004, Kayseri
  - Investigational Site Number : 7920011, Mersin
  - Investigational Site Number : 7920007, Samsun
- United Kingdom (5):
  - Investigational Site Number : 8260003, Portsmouth, Hampshire
  - Investigational Site Number : 8262602, London, London, City of
  - Investigational Site Number : 8262601, London, London, City of
  - Investigational Site Number : 8260006, Glasgow
  - Investigational Site Number : 8260004, Leicester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17560 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25575&tenant=MT_SNY_9011